CLINICAL TRIAL: NCT06726967
Title: The Relationship Between Vitamin D Levels, Thyroid Functions, and Thyroid Autoimmunity
Brief Title: Vitamin D, Hashimato's Thyroiditis and Thyroid Functions
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA005
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Vitamin D; Thyroid Autoimmune Disease
Keywords: vitamin D; Thyroid autoimmunity; hashimato's thyroiditis; thyroid functions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Patients with thyroid function tests (thyroid-stimulating hormone (TSH), free T3 (fT3), free T4 (fT4)), thyroid antibodies (anti-Tg, anti-TPO), and 25(OH) vitamin D levels
  Interventions: Diagnostic Test: vitamin D 25(OH)D

INTERVENTIONS:
Diagnostic Test: vitamin D 25(OH)D — Thyroid functions (thyroid-stimulating hormone (TSH), serbest triiodothyronine (fT3), serbest thyroxine (fT4)); Thyroid antibodies (Anti-thyroid peroxidase (anti-TPO), anti-thyroglobulin (anti-TG))
  Other Names: Thyroid functions; Thyroid antibodies

SUMMARY:
The goal of this retrospective observational study is to determine whether vitamin D levels differ in patients with Hashimoto's thyroiditis (HT) compared to those without Hashimoto's thyroiditis. The main research questions are:

Are vitamin D levels lower in HT patients compared to non-HT patients? Do vitamin D levels vary between HT and non-HT patients based on thyroid function status?

The study was conducted by retrospectively reviewing the medical records of patients who visited the hospital outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following biochemical parameters:

* Vitamin D (25(OH)D) levels
* Thyroid-stimulating hormone (TSH) levels
* Free triiodothyronine (fT3) levels
* Free thyroxine (fT4) levels
* Anti-thyroid peroxidase (anti-TPO) levels
* Anti-thyroglobulin (anti-Tg) levels

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who apply to the Endocrinology Clinic of Ankara Bilkent City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 81180 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D 25 OH D | Baseline
  nmol/L
thyroid-stimulating hormone (TSH) | Baseline
  uIU/mL
free thyroxine (fT4) | Baseline
  ng/dL
Anti-thyroid peroxidase (anti-TPO) | Baseline
  IU/mL
anti-thyroglobulin (anti-TG) | Baseline
  IU/mL

SECONDARY OUTCOMES:
free triiodothyronine (fT3) | Baseline
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Rahime E Karakaya, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)